CLINICAL TRIAL: NCT01120678
Title: Improved Detection of Neonatal Sepsis Using a Targeted Biomarker Assay
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Wallace H. Coulter Foundation (Other)
Responsible Party: Principal Investigator, Karen Fairchild, MD, Professor of Pediatrics, University of Virginia
Other Study IDs: 13987
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Neonatal Sepsis
Keywords: cytokines; neonatal sepsis; diagnosis of sepsis; bacteremia; blood culture; clinical sepsis
MeSH Terms: conditions — Neonatal Sepsis; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples of whole blood were obtained and processed to collect and retain only serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neonates assessed for sepsis.

SUMMARY:
The purpose of this study is to determine whether analysis of specific serum biomarkers will improve the diagnosis of late onset neonatal sepsis and to determine the correlation between plasma levels of specific cytokines and bacteremia in NICU patients >3 days of age.

DETAILED DESCRIPTION:
All infants in the Newborn Intensive Care Unit greater than three days old that had blood cultures sent were eligible for this study. Left-over blood from the time at blood culture was collected for research purposes. Study personnel separated the serum and stored samples at -80 degrees until analysis. Samples were analyzed in batch for neonatal sepsis biomarkers using an antibody-coated microsphere assay with dual laser detection. Clinical information collected included symptoms prompting the blood culture, CBC and culture results, and antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* NICU patients > 3 days of age

Exclusion Criteria:

* less than 3 days old or no waste blood available

Min Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infants in the Newborn Intensive Care Unit greater than three days of age undergoing sepsis evaluation.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cytokine response | Within the first twenty-four hours after blood cultures are obtained.

SECONDARY OUTCOMES:
Heart rate characteristics | Within twenty-fours pre and post blood culture.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fairchild, MD, Principal Investigator — University of Virginia School of Medicine
Locations (2):
- United States (2):
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Virginia Neonatal Intensive Care Unit, Charlottesville, Virginia